CLINICAL TRIAL: NCT06412484
Title: Low Back Pain - Disentangling Trait-Like and State-Like Alterations
Brief Title: State vs. Trait Alterations in Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Schweinhardt Petra (Other)
Responsible Party: Sponsor-Investigator, Schweinhardt Petra, Prof. Dr. Med. PhD, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Other Study IDs: CRPP Renewal
Record Dates: First submitted 2024-01-22; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: Trait vs. State Alterations
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Back Pain (LBP) Patients: LBP patients will undergo three study visits, at moments at which their pain status is different: a) "pain-free", b) low back pain (clinically relevant), c) experimental pain (clinically irrelevant). Measures will be repeated in each visit, to understand the influence / relationship of pain state on possible mechanistic alterations observed in LBP compared to HCs.
  Interventions: Behavioral: Pain Free Session; Behavioral: Low Back Pain Session (= clinically relevant pain); Behavioral: Experimental Pain Session (= clinically irrelevant pain)
- Healthy Controls (HCs): HCs will undergo one single visit, equivalent to patients' "pain-free" visit.
  Interventions: Behavioral: Pain Free Session

INTERVENTIONS:
Behavioral: Pain Free Session — On a day in which participants don't have any pain or a pain ranging from 0-2 (on a numerical rating scale of 0-10), they will undergo all the study measures (see primary outcome measures for detail): clinical exam, QST, SSRs, CPM, rsMRI, lumbar MRI, MRS, and blood sample.
Behavioral: Low Back Pain Session (= clinically relevant pain) — On a day in which patients have an ongoing typical low back pain episode of an intensity of 3 or more (on a numerical rating scale of 0-10), they will undergo all the study measures (see primary outcome measures for detail), except the lumbar MRI: clinical exam, QST, SSRs, CPM, rsMRI, MRS, and blood sample.
  Groups: Low Back Pain (LBP) Patients
Behavioral: Experimental Pain Session (= clinically irrelevant pain) — On a day in which participants don't have any pain or a pain ranging from 0-2 (on a numerical rating scale of 0-10), an experimental pain state will be induced using a high concentration (8%) Qutenza patch, containing capsaicin. All the study measures will be performed (see primary outcome measures for detail), except the lumbar MRI and blood sample: clinical exam, QST, SSRs, CPM, rsMRI, MRS.
  Groups: Low Back Pain (LBP) Patients

SUMMARY:
The primary goal of this study is to investigate whether different alterations observed in patients with non-specific episodic low back pain (compared to healthy volunteers), detected using several assessments: psychophysical and neurophysiological testing, imaging, and blood sampling, are dependent or independent of the presence and type of pain experienced at the time of investigation.

DETAILED DESCRIPTION:
The study consists of three visits (healthy volunteers will only have one pain-free visit), in which patients will be tested in a different "pain state" at each visit:

1. Pain-free visit: will be carried out when the patients have no or little (Numerical Pain Rating Scale (NPRS) </= 2/10) clinical pain.
2. Clinically relevant Low Back Pain visit: will be carried out with patients experiencing a low back pain episode with an intensity of 3/10 or more on the NPRS.
3. Experimental pain / Clinically irrelevant pain visit: will be carried out with the application of a high concentration (8%) Qutenza® capsaicin patch at the arm.

Each of the visits will consist of psychophysical testing, neurophysiological assessement of sweat activity in response to pain, brain resting state magnetic resonance imaging and magnetic resonance spectroscopy. Additionally, and depending on the type of session, a lumbar spine magnetic resonance image (only pain-free session, as characterization) and a blood sample (only pain free and low back pain visit) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* German or English proficiency
* Informed consent
* Low back pain for more than 3 months
* Low back pain clinically not attributable to "red flags" (e.g. infection, fractures, inflammation)
* Fluctuating course of pain (with on and off pain periods).

Exclusion Criteria (applicable to both groups):

* Inability to give informed consent / follow study instructions (e.g. due to language problems)
* Major medical or psychiatric condition. E.g. severe heart disease, diabetes, autoimmune disorders, rheumatic disorders, major depressive disorder, etc.
* Symptomatic radiculopathy, manifested through motor and/or sensory deficits / or signs of nerve root involvement on lumbar MRI.
* Back operation
* BMI > 30
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of people that suffer from non-specific low back pain, meaning that their pain cannot reliably be attributed to a specific pathology and radiographic abnormalities correlate poorly with patients' symptoms.
  Participants should suffer from chronic episodic low back pain, meaning that they have had back pain pain for at least more than 3 months, with recurrent fluctuating pain episodes.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mechanical Detection Threshold (MDT) | 1 - 6 months
  A reduced psychophysical QST battery will be performed in 3 body areas: most painful (MP), adjacent to MP, and a control area.
  MDT will be assessed with Von Frey filaments applied to the skin (mN). Subject reports when tactile input is detected.
Mechanical Pain Threshold (MPT) | 1 - 6 months
  A reduced psychophysical QST battery will be performed in 3 body areas: most painful (MP), adjacent to MP, and a control area.
  MPT will be assessed with pin-pricks (mN) applied to the skin. Subject reports when the stimulus feels sharp or blunt.
Mechanical Pain Sensitivity (MPS) | 1 - 6 months
  A reduced psychophysical QST battery will be performed in 3 body areas: most painful (MP), adjacent to MP, and a control area.
  MPS will be assessed with pin-pricks and Q-tip, cotton swab, and brush applied to the skin. Subjects rate stimuli on scale of 0-100. In our protocol only 3 blocks.
Wind-Up Ratio (WUR) | 1 - 6 months
  A reduced psychophysical QST battery will be performed in 3 body areas: most painful (MP), adjacent to MP, and a control area.
  WUR will be assessed with a pin-prick, which is applied 10 times in 10 seconds. Subjects rate the series on scale of 0-100. In our protocol, only 3 series.
Vibration Detection Threshold (VDT) | 1 - 6 months
  A reduced psychophysical QST battery will be performed in 3 body areas: most painful (MP), adjacent to MP, and a control area.
  VDT will be assessed with a tuning fork applied to a bony prominence. Subject reports when the vibration can't be felt anymore.
Pressure Pain Threshold (PPT): | 1 - 6 months
  A reduced psychophysical QST battery will be performed in 3 body areas: most painful (MP), adjacent to MP, and a control area.
  PPT will be assessed with an algometer (kg), applied to a muscle. Subject reports when pressure becomes painful.
Sympathetic Skin Responses (SSRs) | 1 - 6 months
  Neurophysiological assessement of sweat activity in response to pain will be recorded with cap electrodes located at the hand. Painful heat stimulation will be applied with a thermode of the Pathway Medoc System. A train of 15 heat stimuli, with an inter-stimulus interval of 13-17 seconds, will be applied. The thermode baseline temperature will be 42ºC and during the stimulation the temperature will quickly ramp up to 52 ºC. Subjects are asked to rate the perception of the stimulus using a pain scale of 0-100. This procedure will be done two times: one at the most painful area of the patients, and the corresponding body area in the matched healthy volunteer, and at the volar forearm as a control pain-free area. This readout is a proxy for sympathetic nervous system activity.
Conditioned Pain Modulation (CPM) | 1 - 6 months
  CPM measures the modulation of a noxious test stimulus by another noxious conditioning stimulus applied at a remote body region. In this study, test stimuli of different modalities (pressure, superficial mechanical, heat or electrical stimuli) will be applied at different body regions before and after or before, during and after a cold water bath or neutral water bath (hand immersion) as conditioning stimulus. Changes in test stimuli read-outs (during-before or after-before) will serve as CPM measure. Negative changes represent inhibitory, positive changes facilitatory CPM effects. For all test stimuli read-outs, CPM effects will be expressed as percentage changes. Test stimuli read-outs include: pain ratings on a scale of 0: no pain, to 100: most intense pain; perception thresholds and pain thresholds (in kg for pressure).
Brain resting state Magnetic Resonance Imaging (rsMRI) | 1 - 6 months
  Measure of the brain's spontaneous activity acquired during resting state using a 7T Siemens scanner.
Lumbar Magnetic Resonance Imaging | 1 - 6 months
  Structural resonance image of lumbar spine section acquired using a 3T Siemens scanner.
Brain Magnetic Resonance Spectroscopy (MRS) | 1 - 6 months
  Imaging method that allows the detection of concentration of certain metabolites in the brain. This data will be acquired using a 3T Phillips scanner.
Blood Sample | 1 - 6 months
  Blood sample of approximately 14 ml will be drawn, in a total of 3 tubes: PAXGene blood RNA tube, Serum tube, and K2 EDTA tube. This will allow analysis of inflammatory molecules (i.e. cytokines) and cell concentrations (i.e. immune cells).

SECONDARY OUTCOMES:
Anxiety and Depression | 1 - 6 months
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS). The HADS is a self-report rating scale of 14 items on a 4-point Likert scale (range 0-3), with 7 items for each subscale (anxiety and depression). The total score is the sum of the 14 items, and for each subscale the score is the sum of the respective seven items (ranging from 0-21). Higher score means more anxiety or depression.
Pain Catastrophizing | 1 - 6 months
  Pain catastrophizing will be assessed using questionnaires as for example the Pain Catastrophizing Scale (0-52; higher score meaning more catastrophizing).
Pain Sensitivity | 1 - 6 months
  Pain sensitivity will be assessed using the Pain Sensitivity Questionnaire (PSQ). It consists of 17 items, with an answer range from 0 (not at all painful) to 10 (most severe pain imaginable). The maximum score is 170, where a higher score indicates a higher pain sensitivity.
Pain Self Efficacy | 1 - 6 months
  Pain self efficacy will be assessed using the Pain Self Efficacy Questionnaire (PSEQ). It consists of 10 items, with an answer range from 0 (not at all confident) to 6 (completely confident). The maximum score is 60, where a higher score indicates a higher pain self efficacy / pain coping capacity.
Back Awareness | 1 - 6 months
  Back awareness will be assessed using the Fremantle Back Awareness Questionnaire. It consists of 9 items, with an answer range from 0 (never) to 4 (always). The maximum score is 36, where a higher score indicates a decreased back awareness.
Central sensitization | 1 - 6 months
  Central sensitization symptoms will be assessed using the Central Sensitization Inventory (CSI), which consists of two parts.
  Part A: includes 25 questions assessing typical central sensitisation symptoms. Each answer is scored on a scale of 0 (never) to 4 (always). A score of more than 40 indicates the presence of central sensitisation.
  Part B: determines if the patient has been diagnosed with certain central sensitivity disorder or related disorders, such as anxiety and depression.
Widespread Pain Index (WPI) | 1 - 6 months
  Presence of fibromyalgia symptoms will be assessed using the WPI. In the WPI, patients report body areas in which they have had pain in the past week. Each marked area adds one point, to reach a total score of 19.
  A patient would meet the criteria for fibromyalgia if:
  * WPI score (Part 1) is 7 or higher and SSS score (see below) (Part 2a & b) is 5 or higher OR
  * WPI score (Part 1) is from 3 to 6 AND the SSS score (Part 2a & b) is 9 or higher.
Symptom Severity Scale (SSS) | 1 - 6 months
  Presence of fibromyalgia symptoms will be assessed using the SSS. SSS consists of two parts. In part A patients report the severity of fatigue, waking unrefreshed, and cognitive symptoms. Each question can be answered from 0-3, for a total of 9. The higher the score, the higher the severity of these symptoms. In part B, patients report other somatic symptoms that they have experienced in the past week, reaching a total score of 3. Parts A and B, have a total score of 12 put together.
  A patient would meet the criteria for fibromyalgia if:
  * WPI score (see above) (Part 1) is 7 or higher and SSS score (Part 2a & b) is 5 or higher OR
  * WPI score (Part 1) is from 3 to 6 AND the SSS score (Part 2a & b) is 9 or higher.
Neuropathic Pain | 1 - 6 months
  Neuropathic pain components will be assessed using PainDETECT, which consists of 9 items: 7 weighted sensory descriptor items (never to very strongly) and 2 items relating to spatial and temporal pain characteristics. A score of 19 or more (out of 38) indicates likely neuropathic pain.
Disability | 1 - 6 months
  Patients' functional disability will be measured using the Oswestry Disability Index (ODI), which consists of 10 items addressing different aspects of life (i.e. walking, social life, hygiene, etc.). Each item, has a possible 5 point answer. A higher score indicates higher functional disability.
Pain Extent | 1 - 6 months
  Low back pain patients will be asked to complete pain drawings indicating painful body regions. The painful body area will be calculated as percentage of the whole body area. Higher percentages represent more widespread pain.

CONTACTS AND LOCATIONS:
Overall Officials: Petra Schweinhardt, Principal Investigator — University of Zurich
Locations (1):
- Balgrist Campus, Zurich, Switzerland